CLINICAL TRIAL: NCT03895645
Title: Connors Protocol for the Management and Use of Stored Human Specimens
Brief Title: Connors Protocol for the Management and Use of Stored Human Specimens (Stored Human Specimens)
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999919074; 19-I-N074
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-02

CONDITIONS: Healthy Volunteer Samples
Keywords: Stored Samples; Natural History

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Participants: Participants on the studies' samples that are transferred to this protocol

SUMMARY:
Background:

The HIV research program is part of the National Institute of Allergy and Infectious Diseases. The program aims to learn more about HIV. It also aims to improve the health of people with HIV and create HIV vaccines. People enrolled in prior HIV studies provided samples or data. They consented for their samples or data to be used for future research. Researchers want to keep studying the stored samples and data.

Objective:

To give approved researchers access to stored samples and data after the study of sample origin is over. To do this with human subjects protection oversight by the NIH institutional review board (IRB).

Eligibility:

The study populations were defined by the protocols under which the samples or data were obtained: 11-I-0259, 13-I-0081, and 14-I-0011.

Design:

All participants consented to provide blood or other samples. Their consent included future use of the samples.

Researchers will not contact participants without prior approval of the IRB or the original study protocol.

Samples will be labeled with a code. They will not be labeled with information that identifies the participants.

Participants data will be stored in computers. The computers will be protected with passwords.

This protocol will be kept open as long as the samples or data can be used for future research. When there is no longer a need, the samples may be moved if the IRB approves this. Otherwise they will be destroyed.

...

DETAILED DESCRIPTION:
The HIV intramural research program of NIAID conducts clinical investigations to increase our

knowledge of the biology, pathogenesis and immunology of HIV infection and vaccine

development. After all study-related interventions, follow-up, and primary specimen and data

analyses are complete for an IRB-approved protocol, some human specimens may remain in

storage, and data may continue to be analyzed to meet secondary and exploratory objectives. This protocol will allow for additional laboratory and data analyses to be continued to complete the analyses described under closed NIAID protocol #14-I-0011, Phase 1 Study of Safety and Immunogenicity of Ad4-HIV Vaccine Vectors in Healthy Volunteers.

ELIGIBILITY:
* The study populations were defined by the original protocols under which the stored specimens and/or data were collected. The total population included on this omnibus protocol comprises the

populations of other protocols.

Ages: 18 Years to 116 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Continued analysis | Ongoing
  The objective of this protocol is to continue to have human subjects' protection oversight by the NIH IRB while making stored specimens and/or data available to approved research laboratories and investigators after the study of specimen origin has been terminated. Continued analyses will be for the purpose of research, exploratory immunology, and infectious disease research within the original study objectives and consents under which the specimens and data were collected. Manuscript completion for the primary study objectives will also be covered under this or the original study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Connors, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article after deidentification
Supporting Information: SAP
Time Frame: Immediately following publication
Access Criteria: Anyone who wishes to access the data